CLINICAL TRIAL: NCT06748053
Title: A Multicentre, Randomized, Double-Blind, Placebo Controlled, Dose Finding, Parallel Group, Phase 2 Study of an Anti-TSLP Antibody (GSK5784283) in Adults Aged 18 to 75 Years of Age With Uncontrolled Asthma
Brief Title: A Dose Finding Study With an Anti-TSLP Antibody (GSK5784283) in Adults Aged 18 to 75 Years of Age With Uncontrolled Asthma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 223125; 2024-518321-15 (EudraCT Number)
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Asthma; GSK5784283; Anti-TSLP antibody
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Dose Finding - GSK5784283 (Experimental)
  Interventions: Drug: GSK5784283
- Part A: Dose Finding - Placebo (Experimental)
  Interventions: Drug: Placebo
- Part B: Extended Dosing - GSK5784283 (Experimental)
  Interventions: Drug: GSK5784283
- Part B: Extended Dosing - Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK5784283 — GSK5784283 will be administered.
  Other Names: AIO-001, SHR-1905
  Arms: Part A: Dose Finding - GSK5784283; Part B: Extended Dosing - GSK5784283
Drug: Placebo — Placebo will be administered.
  Arms: Part A: Dose Finding - Placebo; Part B: Extended Dosing - Placebo

SUMMARY:
This study is trying to find the right dose of a long-lasting medicine called GSK5784283 for people with asthma that remains uncontrolled even though they are using regular asthma treatments. GSK5784283 blocks the action of an inflammatory protein called TSLP that may be contributing to your asthma. The study will be conducted in two parts - Part A (dose finding phase) and Part B (extended dosing phase). Part A will assess the lung function, asthma control, participant safety and certain markers of asthma inflammation in the air you breath out and in your blood. Part B will assess the safety and long-term effects of the repeated or single doses of GSK5784283.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Informed Consent: Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol. The participant must be willing and able to comply with trial and follow-up procedures.
* Age: Participants must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
* Documented physician-diagnosed asthma for >= 2 years that meets the National Heart, Lung, and Blood Institute guidelines
* Evidence of variable airflow obstruction consistent with asthma.
* Documented history of asthma exacerbation within 12 months prior to Visit 1.
* An asthma exacerbation defined as a worsening of asthma symptoms.
* A well- documented requirement for regular treatment with medium or high-dose ICS for at least 6 months prior to screening.
* At least one additional maintenance asthma controller medication is required according to standard practice of care (e.g., long-acting beta 2 agonist (LABA), leukotriene receptors antagonists (LTRA), theophylline, long-acting muscarinic antagonist (LAMA), chromones, etc.). Use of additional asthma controller medications must be documented for at least 3 months prior to Visit 1.
* Weight >=40 kg.
* Male or eligible Female.
* Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WONCBP) OR
  * Is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1%, 28 days prior to the 1st dose of the study drug and during the study intervention period and follow-up period. The investigator should evaluate potential for contraceptive method failure (e.g. non-compliance, recently initiated) in relationship to the first dose of study intervention.
  * A WOCBP must have a negative serum pregnancy test at screening and a highly sensitive pregnancy test ([urine or serum] as required by local regulations) within 24 hours before each dose of study intervention.
  * If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
  * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
  * Contraceptive use by women should be consistent with location regulations regarding the methods of highly effective contraception for those participating in clinical trials.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

• Any concomitant respiratory disease that in the opinion of the investigator and/or medical monitor will interfere with the evaluation of the investigational product or interpretation of subject safety or study results (e.g., current upper or lower respiratory tract infection, chronic obstructive pulmonary disease, cystic fibrosis, pulmonary fibrosis, bronchiectasis, allergic bronchopulmonary aspergillosis, Churg-Strauss syndrome, primary ciliary dyskinesia).

Helminth parasitic infection diagnosed within 6 months prior to Visit 1 that has not been treated with, or has failed to respond to, standard of care therapy.

* Active or latent tuberculosis:

  * Participants with a diagnosis or evidence of active or latent tuberculosis are excluded from the study.
  * Diagnosis of vocal cord dysfunction, dysfunctional breathing, or pseudo steroid resistant asthma.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 5 years prior to screening (Participants that had localized carcinoma of the skin which was resected for cure will not be excluded).
* History of an unresolved clinically significant infection within 30 days prior to Visit 1.
* A known immunodeficiency (e.g. human immunodeficiency virus - HIV), other than that explained by the use of corticosteroids taken as therapy for asthma.
* Participants who have known, pre-existing, clinically significant cardiac, endocrine, autoimmune, rheumatologic, metabolic, neurological, renal, gastrointestinal, hepatic, hematological or any other system abnormalities that are uncontrolled with standard treatment including eosinophilic conditions such as hyper-eosinophilic syndrome (HES) and eosinophilic granulomatosis with polyangiitis (EGPA).
* Any clinically relevant abnormal findings in physical examination, hematology, clinical chemistry, urinalysis, vital signs at Visit 2 which in the opinion of the investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to participate in the study.
* Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives prior to Visit 1, whichever is longer and up until the end of study.
* Receipt of any investigational non-biologic agent within 30 days or 5 half-lives prior to screening, whichever is longer and up until the end of study.
* Experimental vaccines are not permitted within 30 days prior to randomization and up until the end of the study.
* Use of immunosuppressive medication (e.g., methotrexate, troleandomycin, oral gold, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, systemic (oral) corticosteroids) within 3 months prior to Visit 1 and up until the end of study.
* Systemic corticosteroid burst including taper within 15 days prior to Visit 1 or during the screening/run-in period.
* Subjects who have not responded to Tezepelumab treatment.
* Receipt of live or live attenuated vaccine(s) within 30 days prior to randomization or plans to receive such vaccines up until the end of study.
* A positive human immunodeficiency virus (HIV) test at screening or subject taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Positive test for hepatitis B virus (HBV) defined as either:

  1. positive for hepatitis B surface antigen (HBsAg) OR
  2. positive for HBV DNA
* Positive Hepatitis C antibody test result.
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* Current smokers (tobacco and marijuana) or former smokers with a smoking history >=10 pack years and subjects using vaping products, including electronic cigarettes.
* History of chronic alcohol or drug abuse within 2 years.
* History of severe allergic reaction, anaphylaxis or documented immune complex disease (Type III hypersensitivity reactions) to any biologic therapy.
* History of sensitivity to any component of the investigational product formulation or a history of drug or other allergy that, in the opinion of the investigator or medical monitor contraindicates their participation.
* Participants who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.
* Participants who meet the following based on results from sample taken at Visit 2:

  1. Alanine aminotransferase (ALT) >2x upper limit of normal (ULN)
  2. Total bilirubin >1.5x ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
  3. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF >= 450 msec or QTcF >= 480 msec for patients with bundle branch block or an abnormal ECG finding that is considered to be clinically significant and would impact the participant's participation during the study, based on the evaluation of the investigator in the 12-Lead ECG central over-read from screening Visit 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
Part A: Change from baseline in the fraction of exhaled nitric oxide (FeNo) | Baseline (Day 1) and at 2, 4, 8,12, 20 and 26 weeks

SECONDARY OUTCOMES:
Part A: Change from baseline in blood eosinophil counts | Baseline (Day 1) and at 2, 4, 8,12, 20 and 26 weeks
Part A: Change from baseline in the forced expiratory volume (FEV1) [pre-and post-bronchodilator | Baseline (Day 1) and at 2, 4, 8,12, 20 and 26 weeks
Part A: Change from baseline in the forced vital capacity (FVC) [pre-and post-bronchodilator | Baseline (Day 1) and at 2, 4, 8,12, 20 and 26 weeks
Part A: Change from baseline in the 5-item Asthma Control Questionnaire (ACQ-5) | Baseline (Day 1) and at 2, 4, 8,12, 20 and 26 weeks
  The ACQ-5 is a five-item questionnaire, which has been developed as a measure of participants' asthma control. The five questions enquire about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, and shortness of breath, wheeze) over the previous week. The response options for all these questions consist of a zero (no impairment/limitation) to six (total impairment/ limitation) scale.
Part A: Maximum Observed Plasma Concentration (Cmax) of GSK5784283 | Up to 26 weeks
Part A: Time to Reach Cmax (Tmax) of GSK5784283 | Up to 26 weeks
Part A: Area under the curve over the dosing interval (AUC0-tau) of GSK5784283 | Up to 26 weeks
Part A & B: Number of participants with treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) | Up to 52 weeks
Part A & B: Number of participants with clinically significant changes in hematology, clinical chemistry and urinalysis | Up to 52 weeks
Part A & B: Number of participants with clinically significant changes in vital signs, including blood pressure, body temperature, and pulse rate | Up to 52 weeks
Part A & B: Number of participants with clinically significant changes in Electrocardiogram (ECG) | Up to 52 weeks
Part A & Part B: Number of participants with treatment-emergent Anti-drug antibodies (ADA) to GSK5784283 | Up to 52 weeks
Part A & Part B: Titers of ADA to GSK5784283 | Up to 52 weeks
Part A: Number of participants with Neutralizing Antibody (NAb) to GSK5784283 | Baseline (Day 1) and at 2, 4, 8,12, 20 and 26 weeks
Part B: Change from baseline in the fraction of exhaled nitric oxide (FeNo) | Baseline (Day 1) and at 2, 4, 8,12, 20, 26, 28, 30, 34, 38, 46, and 52 weeks
Part B: Change from baseline in blood eosinophil counts | Baseline (Day 1) and at 2, 4, 8,12, 20, 26, 28, 30, 34, 38, 46, and 52 weeks
Part B: Ratio to change from baseline in FeNO and blood eosinophil counts | Baseline (Day 1) and 52 weeks
Part B: Change from baseline in the forced expiratory volume (FEV1) [pre-and post-bronchodilator | Baseline (Day 1) and at 2, 4, 8,12, 20, 26, 28, 30, 34, 38, 46, and 52 weeks
Part B: Change from baseline in the forced vital capacity (FVC) [pre-and post-bronchodilator | Baseline (Day 1) and at 2, 4, 8,12, 20, 26, 28, 30, 34, 38, 46, and 52 weeks
Part B: Change from baseline in the 5-item Asthma Control Questionnaire (ACQ-5) | Baseline (Day 1) and at 2, 4, 8,12, 20, 26, 34, 46, and 52
  The ACQ-5 is a five-item questionnaire, which has been developed as a measure of participants' asthma control. The five questions enquire about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, and shortness of breath, wheeze) over the previous week. The response options for all these questions consist of a zero (no impairment/limitation) to six (total impairment/ limitation) scale.
Part B: Number of participants with Neutralizing Antibody (NAb) to GSK5784283 | Baseline (Day 1) and at 2, 4, 8,12, 20, 26, 28, 30, 34, 38, 46, and 52 weeks

CONTACTS AND LOCATIONS:
Locations (116):
- United States (50):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Redding, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Leesburg, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Sanford, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Lathrup Village, Michigan
  - GSK Investigational Site, Warren, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Pineville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, DuBois, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Cypress, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, American Fork, Utah
  - GSK Investigational Site, Pleasant View, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Ogden, Utah
  - GSK Investigational Site, Bellingham, Washington
- Bulgaria (10):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Gorna Oryahovitsa
  - GSK Investigational Site, Lovech
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Vratsa
- Canada (6):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (3):
  - GSK Investigational Site, Brandýs nad Labem
  - GSK Investigational Site, Mladá Boleslav
  - GSK Investigational Site, Teplice
- Germany (11):
  - GSK Investigational Site, Bendorf
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Darmstadt
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Fürstenwalde
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Magdeburg
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, München
  - GSK Investigational Site, Neu-Isenburg
  - GSK Investigational Site, Schleswig
- Japan (17):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yokohama
- Romania (6):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova Dolj
  - GSK Investigational Site, Timișoara
- Spain (10):
  - GSK Investigational Site, Alcorcon Madrid
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benalmádena
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- United Kingdom (3):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/